CLINICAL TRIAL: NCT00240682
Title: Phase II Study of Cetuximab as Monotherapy and First Line Treatment in Patients With Locally Advanced or Metastatic Squamous Cell Carcinoma of the Skin Expressing EGFR.
Brief Title: Study of Cetuximab in Squamous Cell Carcinoma of the Skin Expressing EGFR
Acronym: CTXSCC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Hospitalier of Chartres (Other)
Collaborators: Hospital of Chartres- France (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2005-001098-82
Record Dates: First submitted 2005-10-17; First posted 2005-10-18 (Estimated); Last update posted 2012-02-22 (Estimated); Status verified 2009-08

CONDITIONS: Skin Diseases; Carcinoma, Squamous Cell
Keywords: Carcinoma, Squamous Cell; Skin; cetuximab; epidermal growth factor receptor
MeSH Terms: conditions — Skin Diseases; Carcinoma, Squamous Cell | interventions — Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- cetuximab (Experimental): cetuximab
  Interventions: Drug: cetuximab

INTERVENTIONS:
Drug: cetuximab — Dosage form: bottles of 50 ml, 2 mg/ml; Dosage:400 mg/m2 initial dose followed by 250 mg/m2 by infusion every week; Number of Cycles : until progression or unacceptable toxicity develops.
  Other Names: Erbitux

SUMMARY:
The purpose of this study is to determine whether cetuximab is effective in the treatment of locally advanced or metastatic squamous cell carcinoma of the skin expressing EGFR.

DETAILED DESCRIPTION:
Patients with locally advanced or metastatic squamous cell carcinoma (SCC) of the skin are often bad responders to conventional chemotherapy included cisplatin.

The investigation of the EGFR expression may allow identifying new molecular targets for novel therapeutic strategies in patients with locally advanced or metastatic SCC of the skin.

Several publications in the literature for primary lesions and one publication for metastatic lesions showed that EGFR was expressed in 80-90% of SCC of the skin. Immunohistochemistry studies performed at the Gustave Roussy Institute confirm these data: they found an over-expression of EGFR in 90% of patients with metastatic disease. These results are in favor of the investigation of cetuximab in patients with locally advanced or metastatic SCC of the skin expressing EGFR.

Cetuximab is a monoclonal antibody targeted against EGFR administered weekly by intravenous route; it may be prescribed as out hospital to patients with locally advanced or metastatic SCC of the skin expressing EGFR.

Due to the low occurrence of locally advanced or metastatic SCC of the skin, a multicenter trial will be required.

ELIGIBILITY:
Inclusion Criteria:

* Histological SCC of the skin expressing (IHC) moderately or highly the EGFR (++ and +++, on a semi-quantitative scale).
* Locally advanced or metastatic SCC of the skin not suitable for local surgery with documented progression.
* Presence of at least one measurable target lesion by RECIST criteria.
* At least one lesion accessible to biopsies.
* ECOG Performance status < 2.
* Life expectancy > 3 months.
* Age > 18 years.
* Normal hematological (Neutrophils > 1.5x109 cells/l, platelets > 100x109 cells/l), hepatic (bilirubin < 1.5 times the upper limit of the normal range (ULN); alkaline phosphatase and transaminases < 5 x UNL in case of hepatic metastases or < 2.5 x UNL in absence of hepatic metastases) and renal (serum creatinine < 150 micromol/L) functions.
* Written informed consent.
* In case of second tumor,excepted carcinoma of the cervix and adequately treated basal or squamous cell skin carcinoma, the possibility for including a patient may be discussed with the principal investigator.

Exclusion Criteria:

* Prior chemotherapy
* Prior radiotherapy < 1 month.
* Prior therapy with agent targeting EGFR
* Unstable systemic diseases or active uncontrolled infections.
* Patients (male and female) not using effective contraception if of reproductive potential.
* Females pregnant or lactating. Women of child bearing potential must have a negative serum or urine pregnancy test prior to start each cycle of treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2005-10; Primary Completion 2009-04 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Disease control rate assessed by CT or MRI | 6 weeks

SECONDARY OUTCOMES:
Safety profile. | during treatment or within 30 days after the final administration with a cut-off date at week 48.
Time to disease progression. | number of days from the start of treatment to the earliest day of progressive disease
Overall survival. | from the first infusion until week 48 or death
Duration of response in responder patients at 6 weeks. | time to disease progression

CONTACTS AND LOCATIONS:
Overall Officials: Eve Maubec, MD, Principal Investigator — Dermatology Department, Hospital Bichat, Paris, France
Locations (14):
- France (14):
  - Hospital of Caen, Caen
  - Hospital of Chartres, Chartres
  - Hospital Hôtel Dieu, Clermont-Ferrand
  - Beaujon's Hospital, Clichy
  - CHR of Colmar, Colmar
  - Hospital Henri Mondor, Créteil
  - Hospital Tarnier-Cochin, Paris
  - Hospital Saint Louis, Department of P. Morel, Paris
  - Hospital Saint-Louis, department of L. Dubertret, Paris
  - Hospital Bichat, Paris
  - Hospital of Reims, Reims
  - Hospital Pontchaillou, Rennes
  - Eugène Marquis Center, Rennes
  - Hospital Charles Nicolle, Rouen

REFERENCES:
- [Background] Maubec E, Duvillard P, Velasco V, Crickx B, Avril MF. Immunohistochemical analysis of EGFR and HER-2 in patients with metastatic squamous cell carcinoma of the skin. Anticancer Res. 2005 Mar-Apr;25(2B):1205-10. PMID 15865067
- [Background] Alam M, Ratner D. Cutaneous squamous-cell carcinoma. N Engl J Med. 2001 Mar 29;344(13):975-83. doi: 10.1056/NEJM200103293441306. No abstract available. PMID 11274625
- [Background] Shimizu T, Izumi H, Oga A, Furumoto H, Murakami T, Ofuji R, Muto M, Sasaki K. Epidermal growth factor receptor overexpression and genetic aberrations in metastatic squamous-cell carcinoma of the skin. Dermatology. 2001;202(3):203-6. doi: 10.1159/000051637. PMID 11385224
- [Background] Huang SM, Bock JM, Harari PM. Epidermal growth factor receptor blockade with C225 modulates proliferation, apoptosis, and radiosensitivity in squamous cell carcinomas of the head and neck. Cancer Res. 1999 Apr 15;59(8):1935-40. PMID 10213503
- [Background] Barbara A Burtness, Yi Li, William Flood, Bassam I Mattar, Arlene A Forastiere. Phase III trial comparing cisplatin (C) + placebo (P) to C + anti-epidermal growth factor antibody (EGF-R) C225 in patients (pts) with metastatic/recurrent head & neck cancer (HNC). Journal of Clinical Oncology,2002 ASCO Annual Meeting Proceedings. Abstract 901.
- [Background] Nemunaitis JJ, Eiseman I, Cunningham C et al. A phase I trial of CI-1033, a pan-erbB tyrosine kinase inhibitor, given daily for 14 days every 3 weeks, in patients with advanced solid tumors. Proc Am Soc Clin Oncol 22: page 243, 2003 (abstr 974).
- [Result] Maubec E, Petrow P, Scheer-Senyarich I, Duvillard P, Lacroix L, Gelly J, Certain A, Duval X, Crickx B, Buffard V, Basset-Seguin N, Saez P, Duval-Modeste AB, Adamski H, Mansard S, Grange F, Dompmartin A, Faivre S, Mentre F, Avril MF. Phase II study of cetuximab as first-line single-drug therapy in patients with unresectable squamous cell carcinoma of the skin. J Clin Oncol. 2011 Sep 1;29(25):3419-26. doi: 10.1200/JCO.2010.34.1735. Epub 2011 Aug 1. PMID 21810686